CLINICAL TRIAL: NCT04378569
Title: A Phase 1/2b, Multiple Dose and 12-Week, Parallel Group, Double Blind, Dose Ranging, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-252 Cream 0.1% and ARQ-252 Cream 0.3% in Subjects With Chronic Hand Eczema
Brief Title: Safety and Efficacy of ARQ-252 Cream in Subjects With Chronic Hand Eczema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ-252-205
Record Dates: First submitted 2020-04-30; First posted 2020-05-07 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Chronic Hand Eczema

STUDY DESIGN:
Intervention Model Description: There are 2 cohorts of subjects.
  * Cohort 1 (Phase 1) is a multiple dose cohort in which subjects with chronic hand eczema will be assigned to ARQ-252 cream 0.3% QD x 2 weeks to be applied to both hands (approximately 4% of BSA).
  * Cohort 2 (Phase 2b) is a parallel group, double blind, vehicle-controlled cohort in which subjects with chronic hand eczema will be randomized to ARQ-252 cream 0.3% QD, ARQ-252 cream 0.3% BID, ARQ-252 cream 0.1% QD, vehicle cream BID or vehicle cream QD x 12 weeks to be applied to both hands (approximately 4% of BSA).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ARQ-252 cream 0.3% QD (once daily) (Active Comparator): Active Comparator
  Interventions: Drug: ARQ-252 cream 0.3%
- ARQ-252 cream 0.3% BID (twice daily) (Active Comparator): Active Comparator
  Interventions: Drug: ARQ-252 cream 0.3%
- ARQ-252 cream 0.1% QD (once daily) (Active Comparator): Active Comparator
  Interventions: Drug: ARQ-252 cream 0.1%
- Vehicle cream BID (twice daily) (Placebo Comparator): Placebo Comparator
  Interventions: Drug: ARQ-252 Vehicle Cream
- Vehicle cream QD (once daily) (Placebo Comparator): Placebo Comparator
  Interventions: Drug: ARQ-252 Vehicle Cream

INTERVENTIONS:
Drug: ARQ-252 cream 0.3% — ARQ-252 cream 0.3%
  Arms: ARQ-252 cream 0.3% BID (twice daily); ARQ-252 cream 0.3% QD (once daily)
Drug: ARQ-252 cream 0.1% — ARQ-252 cream 0.1%
  Arms: ARQ-252 cream 0.1% QD (once daily)
Drug: ARQ-252 Vehicle Cream — ARQ-252 Vehicle Cream
  Arms: Vehicle cream BID (twice daily); Vehicle cream QD (once daily)

SUMMARY:
This study will assess the safety and efficacy of ARQ-252 cream in subjects with chronic hand eczema

DETAILED DESCRIPTION:
This is a Phase 1/2b multiple dose, parallel group, double blind, vehicle-controlled study of the safety and efficacy of ARQ-252 cream in subjects with chronic hand eczema

ELIGIBILITY:
Inclusion Criteria

* Participants legally competent to sign and give informed consent.
* Males and females 18 years of age and older (inclusive) at the time of consent.
* Clinical diagnosis of chronic hand eczema, defined as hand eczema persistent for more than 3 months, or returned twice or more within the last 12 months. Generally stable disease for 6 weeks.
* Chronic hand eczema involving at least 0.3% body surface area total (i.e., approximately a third of one handprint) lesions on both hands added together
* Female subjects of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Baseline. For FOCBP involved in any sexual intercourse that could lead to pregnancy: the subject must agree to use a highly effective contraceptive method for at least 4 weeks prior to Day 1. Additionally, from Day 1 until at least 4 weeks after the last investigational product administration, these subjects must agree to use at least 1 highly effective contraceptive method in addition to 1 barrier method according to the Contraception Requirements Section of the protocol.
* Females of non-childbearing potential must either be post-menopausal with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization.
* Males, if engaging in sexual intercourse with a female who is pregnant or a female of childbearing potential, must agree to use a condom every time during the study and every and every time subsequently until 4 weeks after the last dose of investigational product.
* Subjects in good health as judged by the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry labs, hematology values, and urinalysis.

Exclusion Criteria

* Concurrent skin diseases on the hands which, in the opinion of the Investigator, could confound the study (e.g., tinnea manuum).
* Subjects with any presence or history of psoriasis.
* History of a positive patch test with continued exposure to allergen. Subjects must have undergone diagnostic patch testing within 3 years prior to Baseline (Visit 2).
* Subjects who cannot discontinue systemic and/or topical therapies for the treatment of chronic hand eczema prior to Baseline and during the study
* Subjects with a history of chronic alcohol or drug abuse within 6 months prior to Baseline
* Pregnant or lactating women or women planning to become pregnant during the study and / or within 28 days following the last dose of investigational product.
* Subjects with any serious medical condition or clinically significant laboratory, ECG, vital signs or physical examination abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (37):
- United States (25):
  - Arcutis Clinical Site 239, Beverly Hills, California
  - Arcutis Clinical Site 225, Encino, California
  - Arcutis Clinical Site 112, Fremont, California
  - Arcutis Clinical Site 120, Irvine, California
  - Arcutis Clinical Site 208, Santa Monica, California
  - Arcutis Clinical Site 174, Aventura, Florida
  - Arcutis Clinical Site 167, Coral Gables, Florida
  - Arcutis Clinical Site 104, Sanford, Florida
  - Arcutis Clinical Site 214, Indianapolis, Indiana
  - Arcutis Clinical Site 217, Louisville, Kentucky
  - Arcutis Clinical Site 213, Metairie, Louisiana
  - Arcutis Clinical Site 125, Rockville, Maryland
  - Arcutis Clinical Site 212, Detroit, Michigan
  - Arcutis Clinical Site 216, New Brighton, Minnesota
  - Arcutis Clinical Site 171, New York, New York
  - Arcutis Clinical Site 115, High Point, North Carolina
  - Arcutis Clinical Site 173, Portland, Oregon
  - Arcutis Clinical Site 135, Pittsburgh, Pennsylvania
  - Arcutis Clinical Site 162, Austin, Texas
  - Arcutis Clinical Site 104, College Station, Texas
  - Arcutis Clinical Site 164, Houston, Texas
  - Arcutis Clinical Site 163, Pflugerville, Texas
  - Arcutis Clinical Site 161, San Antonio, Texas
  - Arcutis Clinical Site 110, San Antonio, Texas
  - Arcutis Clinical Site 169, Norfolk, Virginia
- Australia (2):
  - Arcutis Clinical Site 306, Westmead, New South Wales
  - Arcutis Clinical Site 303, East Melbourne, Victoria
- Canada (10):
  - Arcutis Clinical Site 207, Surrey, British Columbia
  - Arcutis Clinical Site 205, Ajax, Ontario
  - Arcutis Clinical Site 218, Barrie, Ontario
  - Arcutis Clinical Site 103, London, Ontario
  - Arcutis Clinical Site 133, Mississauga, Ontario
  - Arcutis Clinical Site 165, Oakville, Ontario
  - Arcutis Clinical Site 109, Peterborough, Ontario
  - Arcutis Clinical Site 241, Richmond Hill, Ontario
  - Arcutis Clinical Site 106, Waterloo, Ontario
  - Arcutis Clinical Site 242, Montreal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 36 centers in the United States, Canada, and Australia.
Groups:
- Cohort 1: ARQ-252 Cream 0.3% QD: Participants applied ARQ-252 cream 0.3% QD to both hands for 2 weeks.
- Cohort 2: ARQ-252 Cream 0.3% QD: Participants applied ARQ-252 cream 0.3% QD to both hands for 12 weeks.
- Cohort 2: ARQ-252 Cream 0.3% BID: Participants applied ARQ-252 cream 0.3% BID to both hands for 12 weeks.
- Cohort 2: ARQ-252 Cream 0.1% QD: Participants applied ARQ-252 cream 0.1% QD to both hands for 12 weeks.
- Cohort 2: Vehicle Cream QD: Participants applied ARQ-252 Vehicle Cream QD to both hands for 12 weeks.
- Cohort 2: Vehicle Cream BID: Participants applied ARQ-252 Vehicle Cream BID to both hands for 12 weeks.
Period: Overall Study
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
Started | 7 | 65 | 61 | 32 | 33 | 32
Completed | 7 | 56 | 50 | 28 | 23 | 22
Not Completed | 0 | 9 | 11 | 4 | 10 | 10
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 3 | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 7 | 4 | 5 | 4
Not completed — Lack of response | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID | Total
Number analyzed (Participants) | 7 | 65 | 61 | 32 | 33 | 32 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.18) | 41.6 (15.08) | 43.3 (15.05) | 41.6 (15.33) | 40.3 (12.06) | 43.3 (13.36) | 42.2 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 37 | 39 | 21 | 15 | 23 | 140
  Male | 2 | 28 | 22 | 11 | 18 | 9 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 11 | 12 | 5 | 8 | 5 | 44
  Not Hispanic or Latino | 4 | 54 | 49 | 27 | 25 | 27 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 2 | 3 | 3 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 9 | 8 | 3 | 3 | 4 | 28
  White | 6 | 51 | 48 | 23 | 27 | 25 | 180
  More than one race | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 0 | 0 | 3
Investigator Global Assessment (IGA) Categorical Scores at Baseline [Count of Participants; unit: Participants] — The IGA is 5-point scale assessing the severity of hand eczema; scores range from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity.
  Participants
    0 - Clear | 0 | 0 | 0 | 0 | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0 | 0 | 0 | 0 | 0
    2 - Mild | 1 | 12 | 8 | 8 | 7 | 9 | 45
    3 - Moderate | 5 | 45 | 44 | 21 | 21 | 21 | 157
    4 - Severe | 1 | 8 | 9 | 3 | 5 | 2 | 28
IGA Mean Scores at Baseline [Mean (Standard Deviation); unit: score on a scale] — The IGA is 5-point scale assessing the severity of hand eczema; scores range from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity.
  score on a scale | 3.0 (0.58) | 2.9 (0.56) | 3.0 (0.53) | 2.8 (0.57) | 2.9 (0.61) | 2.8 (0.55) | 2.9 (0.56)
Worst Itch Numerical Rating Scale (WI-NRS) Baseline Score [Mean (Standard Deviation); unit: score on a scale] — The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours (higher scores indicate higher itch severity). Population: All participants with baseline data available are included.
  score on a scale
    number analyzed (Participants) | 7 | 64 | 60 | 32 | 33 | 31 | 227
    (all) | 6.7 (2.56) | 5.8 (2.45) | 5.8 (2.75) | 6.0 (3.19) | 5.5 (2.83) | 5.0 (2.80) | 5.7 (2.74)
Hand Eczema Severity Index (HECSI) Mean Baseline Score [Mean (Standard Deviation); unit: score on a scale] — The HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) on 5 areas of the hand (fingertips, fingers [except tips], palm, back of hand, wrists) by use of a standard scale. Each subscale is scored from 0 to 60; the total HECSI score ranges from 0 to 360 with higher scores indicating greater symptom severity.
  score on a scale | 57.4 (58.35) | 43.7 (31.43) | 43.9 (35.74) | 37.1 (34.51) | 45.8 (50.31) | 38.9 (32.72) | 42.9 (37.08)

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Participants With ≥1 Adverse Event (AE)
Description: The number of Cohort 1 participants with an AE is reported. An AE is any untoward or unfavorable medical occurrence in a human participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to participation in the research.
Time Frame: Up to 3 weeks
Population: All treated participants in Cohort 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 0
Participants | 1 |  |  |  |  |

2. Primary Outcome: Cohort 1: Number of Participants With an Application Site Reaction
Description: The number of Cohort 1 participants with AEs coded as application site events is reported.
Time Frame: Up to 3 weeks
Population: All treated participants in Cohort 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 0
Participants | 0 |  |  |  |  |

3. Primary Outcome: Cohort 1: Number of Participants With ≥1 Serious Adverse Event (SAE)
Description: The number of Cohort 1 participants with an SAE is reported. An SAE is any AE that results in death, is life-threatening (places the subject at immediate risk of death from the event as it occurred), requires inpatient hospitalization or prolongation of existing hospitalization, results in a persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is any other adverse event that, based upon appropriate medical judgment, may jeopardize the subject's health.
Time Frame: Up to 3 weeks
Population: All treated participants in Cohort 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 0
Participants | 0 |  |  |  |  |

4. Primary Outcome: Cohort 1: Number of Participants With Significant Changes in Hematology Laboratory Parameters
Description: The number of Cohort 1 participants with a significant change in hematology is reported.
Time Frame: Up to 3 weeks
Population: All treated participants in Cohort 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 0
Participants | 0 |  |  |  |  |

5. Primary Outcome: Cohort 1: Number of Participants With Significant Changes in Chemistry Laboratory Parameters
Description: The number of Cohort 1 participants with a significant change in chemistry is reported.
Time Frame: Up to 3 weeks
Population: All treated participants in Cohort 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 0
Participants | 0 |  |  |  |  |

6. Primary Outcome: Cohort 2: Investigator's Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 12
Description: The IGA is 5-point scale assessing the severity of hand eczema; scores range from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity. The number of participants with an IGA score of 'clear' or 'almost clear' at Week 12 is presented.
Time Frame: Week 12
Population: Participants from Cohort 2 with data available are included. Note that all Cohort 2 Vehicle Cream (QD or BID) participants are pooled for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Vehicle Cream (Pooled): Participants applied ARQ-252 Vehicle Cream QD or BID to both hands for 12 weeks.
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream (Pooled)
Number analyzed (Participants) | 0 | 59 | 50 | 28 | 46
Participants | 0 | 23 | 15 | 10 | 16
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream (Pooled); Test type: Superiority; p = 0.5788, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score with multiple imputation used to handle missing data; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.49 to 2.53] — Stratified by pooled site group and baseline IGA score with multiple imputation used to handle missing data
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream (Pooled); Test type: Superiority; p = 0.6488, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score with multiple imputation used to handle missing data; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.33 to 2.17] — Stratified by pooled site group and baseline IGA score with multiple imputation used to handle missing data
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream (Pooled); Test type: Superiority; p = 0.5653, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score with multiple imputation used to handle missing data; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.32 to 2.25] — Stratified by pooled site group and baseline IGA score with multiple imputation used to handle missing data

7. Secondary Outcome: Cohort 2: Achievement of IGA Score of 'Clear' or 'Almost Clear' PLUS at Least a 2-point Improvement From Baseline
Description: The IGA is 5-point scale assessing the severity of hand eczema, with scores ranging from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity. The number of participants with an IGA score of 'clear' or 'almost clear' plus ≥2-point improvement (ie, decrease) from Baseline is presented.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Vehicle Cream Pooled: Participants applied ARQ-252 Vehicle Cream QD or BID to both hands for 12 weeks.
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 62 | 58 | 31 | 64
Participants
  Week 2 | 0 | 8 | 6 | 2 | 7
  Week 4: number analyzed (Participants) | 0 | 61 | 56 | 29 | 55
  Week 4 | 0 | 14 | 11 | 2 | 13
  Week 8: number analyzed (Participants) | 0 | 56 | 53 | 27 | 51
  Week 8 | 0 | 12 | 15 | 4 | 14
  Week 12: number analyzed (Participants) | 0 | 59 | 50 | 28 | 46
  Week 12 | 0 | 20 | 13 | 5 | 12
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p = 0.5033, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score with multiple imputation to handle missing data; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.25 to 2.78] — Stratified by pooled site group and baseline IGA score with multiple imputation to handle missing data
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p = 0.4975, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score with multiple imputation to handle missing data; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.25 to 2.79] — Stratified by pooled site group and baseline IGA score with multiple imputation to handle missing data
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; Cochran-Mantel-Haenszel — P value was not evaluable; Stratified by pooled site group and baseline IGA score with multiple imputation to handle missing data; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.04 to 2.55] — Stratified by pooled site group and baseline IGA score with multiple imputation to handle missing data

8. Secondary Outcome: Cohort 2: Achievement of at Least a 2-point Improvement in IGA Score From Baseline
Description: The IGA is 5-point scale assessing the severity of hand eczema, with scores ranging from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity. The number of participants with ≥2-point improvement from baseline in IGA score is presented.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 62 | 58 | 31 | 64
Participants
  Week 2 |  | 9 | 6 | 3 | 9
  Week 4: number analyzed (Participants) | 0 | 61 | 56 | 29 | 55
  Week 4 |  | 15 | 14 | 2 | 13
  Week 8: number analyzed (Participants) | 0 | 56 | 53 | 27 | 51
  Week 8 |  | 13 | 17 | 4 | 14
  Week 12: number analyzed (Participants) | 0 | 59 | 50 | 28 | 46
  Week 12 |  | 22 | 16 | 5 | 13
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p = 0.7237, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.23 to 2.44] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p = 0.8380, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.17 to 2.10] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p-value was unevaluable; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.04 to 2.55] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data

9. Secondary Outcome: Cohort 2: Achievement of IGA Score of 'Clear' or 'Almost Clear'
Description: The IGA is 5-point scale assessing the severity of hand eczema, with scores ranging from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity. The number of participants with ≥2-point improvement from baseline is presented.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 62 | 58 | 31 | 64
Participants
  Week 2 |  | 9 | 7 | 3 | 7
  Week 4 |  | 15 | 13 | 4 | 15
  Week 8 |  | 15 | 16 | 6 | 17
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.9604, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.31 to 3.07] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.9752, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.32 to 3.25] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.5077, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.11 to 3.03] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 4: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.5916, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.26 to 2.15] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 5: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.3320, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.27 to 1.57] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 6: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.1922, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.14 to 1.57] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 7: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.4188, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.23 to 1.81] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 8: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.5520, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.29 to 1.92] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data
Statistical Analysis 9: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.69, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.21 to 2.20] — Stratified by pooled site group and baseline IGA score, with multiple imputation of missing data

10. Secondary Outcome: Cohort 2: Change From Baseline in Investigator's Global Assessment (IGA) Score
Description: The IGA is 5-point scale assessing the severity of hand eczema, with scores ranging from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity. The mean change from baseline in IGA score is presented, with lower scores indicating a reduction in symptom severity.
Time Frame: Weeks 2, 4, 8, and 12
Population: All participants in Cohort 2 are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 65 | 61 | 32 | 65
units on a scale
  Week 2 |  | -0.55 (0.107) | -0.50 (0.109) | -0.35 (0.143) | -0.48 (0.105)
  Week 4 |  | -0.68 (0.126) | -0.71 (0.129) | -0.58 (0.174) | -0.72 (0.129)
  Week 8 |  | -0.73 (0.149) | -0.84 (0.153) | -0.57 (0.203) | -0.78 (0.150)
  Week 12 |  | -1.04 (0.149) | -0.93 (0.155) | -0.73 (0.205) | -0.80 (0.150)
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority — Week 2; p = 0.6464, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables, with multiple imputation of missing data; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.33 to 0.21] — Treatment group, pooled site group, and baseline IGA were independent variables, with multiple imputation of missing data
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.8881, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.29 to 0.25] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.4360, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.20 to 0.46] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.8196, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.29 to 0.36] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.9217, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.31 to 0.34] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p = 0.4783, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.25 to 0.53] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 7: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.7725, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.32 to 0.43] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 8: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.7861, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.43 to 0.33] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 9: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.3521, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.24 to 0.68] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 10: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.2166, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.62 to 0.14] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 11: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.5262, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.52 to 0.27] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 12: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.7575, ANCOVA; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.39 to 0.54] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Cohort 2: Change From Baseline in Worst Itch Numeric Rating Scale (WI-NRS) Score
Description: The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. The mean change from baseline in WI-NRS is reported.
Time Frame: Weeks 2, 4, 8, and 12
Population: All participants in Cohort 2 with data available are included.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 61 | 59 | 32 | 59
score on a scale
  Week 2 |  | -2.43 (0.365) | -2.25 (0.360) | -3.16 (0.469) | -1.80 (0.355)
  Week 4: number analyzed (Participants) | 0 | 60 | 55 | 29 | 54
  Week 4 |  | -3.00 (0.359) | -2.48 (0.372) | -3.75 (0.504) | -2.49 (0.373)
  Week 8: number analyzed (Participants) | 0 | 59 | 51 | 28 | 49
  Week 8 |  | -3.39 (0.338) | -2.85 (0.361) | -3.48 (0.476) | -2.64 (0.362)
  Week 12: number analyzed (Participants) | 0 | 56 | 47 | 28 | 43
  Week 12 |  | -3.71 (0.323) | -3.39 (0.349) | -3.87 (0.444) | -3.08 (0.354)

12. Secondary Outcome: Cohort 2: Achievement of ≥4-point Reduction From Baseline in Worst Itch Numeric Rating Scale (WI-NRS) Pruritus Score
Description: The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours (higher scores indicate higher itch severity). The mean change from baseline in WI-NRS is reported. The number of participants with a baseline WI-NRS score of ≥4 who achieved a ≥4-point reduction is reported.
Time Frame: Weeks 2, 4, 8, and 12
Population: All randomized participants in Cohort 2 with data available and who had baseline WI-NRS scores ≥4 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 48 | 47 | 24 | 42
Participants
  Week 2 |  | 21 | 20 | 14 | 12
  Week 4: number analyzed (Participants) | 0 | 47 | 44 | 21 | 38
  Week 4 |  | 23 | 19 | 15 | 14
  Week 8: number analyzed (Participants) | 0 | 46 | 40 | 20 | 34
  Week 8 |  | 29 | 20 | 15 | 15
  Week 12: number analyzed (Participants) | 0 | 44 | 36 | 20 | 29
  Week 12 |  | 30 | 21 | 16 | 16
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.2662, Cochran-Mantel-Haenszel; Stratified; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.64 to 4.70] — Stratified
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.3798, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.59 to 4.00]
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.0611, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.18, 95% CI 2-sided [0.90 to 11.17]
Statistical Analysis 4: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.3129, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.64 to 3.93]
Statistical Analysis 5: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.9586, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.35 to 2.74]
Statistical Analysis 6: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.0643, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.65, 95% CI 2-sided [0.87 to 15.29]
Statistical Analysis 7: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.0932, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.84 to 6.88]
Statistical Analysis 8: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.5730, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.44 to 4.59]
Statistical Analysis 9: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.0389, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.96, 95% CI 2-sided [0.96 to 25.66]
Statistical Analysis 10: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.2813, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.60 to 5.53]
Statistical Analysis 11: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.6841, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.17 to 3.03]
Statistical Analysis 12: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.3113, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.49 to 9.21]

13. Secondary Outcome: Cohort 2: Change From Baseline in Hand Eczema Severity Index (HECSI) Score
Description: The HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) on 5 areas of the hand (fingertips, fingers [except tips], palm, back of hand, wrists) by use of a standard scale. Each subscale is scored from 0 to 60; the total HECSI score ranges from 0 to 360 with higher scores indicating greater symptom severity. The mean change from baseline in HECSI is reported.
Time Frame: Weeks 2, 4, 8, and 12
Population: All participants in Cohort 2 with data available are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 62 | 58 | 31 | 64
score on a scale
  Week 2 |  | -18.3 (27.39) | -13.6 (21.67) | -4.0 (22.37) | -12.4 (31.84)
  Week 4: number analyzed (Participants) | 0 | 61 | 56 | 29 | 55
  Week 4 |  | -21.3 (28.38) | -21.0 (24.78) | -8.8 (20.22) | -14.6 (30.89)
  Week 8: number analyzed (Participants) | 0 | 56 | 53 | 29 | 55
  Week 8 |  | -22.7 (29.50) | -19.7 (27.12) | -8.3 (25.16) | -17.8 (33.15)
  Week 12: number analyzed (Participants) | 0 | 59 | 50 | 28 | 46
  Week 12 |  | -25.8 (30.25) | -26.3 (29.85) | -14.5 (19.19) | -18.6 (36.12)

14. Secondary Outcome: Cohort 2: Change From Baseline in Numerical Rating Scale (NRS) for Pain Score
Description: The NRS Pain Scale is a widely-used instrument for pain screening. Participants rate the intensity of pain experienced in the past 24 hours on a scale from 0 ('no pain at all') to 10 ('worst pain possible'). The mean change from baseline NRS Pain score is reported.
Time Frame: Weeks 2, 4, 8, and 12
Population: All participants in Cohort 2 with data available are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 62 | 59 | 32 | 58
score on a scale
  Week 2 |  | -1.75 (2.368) | -1.74 (2.464) | -1.86 (2.923) | -0.71 (2.298)
  Week 4: number analyzed (Participants) | 0 | 61 | 56 | 29 | 53
  Week 4 |  | -2.18 (2.611) | -1.66 (2.704) | -2.34 (2.897) | -0.88 (2.176)
  Week 8: number analyzed (Participants) | 0 | 60 | 52 | 28 | 48
  Week 8 |  | -2.15 (2.722) | -1.64 (3.062) | -2.29 (3.224) | -0.89 (2.205)
  Week 12: number analyzed (Participants) | 0 | 57 | 49 | 28 | 42
  Week 12 |  | -2.58 (2.700) | -1.95 (2.708) | -2.11 (3.439) | -1.06 (2.602)

15. Secondary Outcome: Cohort 2: The Rate of Achievement of ≥4-point Reduction From Baseline in Pain Numerical Rating Scale (NRS) Score
Description: The NRS Pain Scale is a widely-used instrument for pain screening. Participants rate the intensity of pain experienced in the past 24 hours on a scale from 0 ('no pain at all') to 10 ('worst pain possible'). The number of participants with ≥4-point reduction from baseline NRS Pain score is reported.
Time Frame: Weeks 2, 4, 8, and 12
Population: All participants in Cohort 2 who had baseline NRS Pain scores ≥4 and with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 30 | 25 | 17 | 20
Participants
  Week 2 |  | 15 | 8 | 8 | 3
  Week 4: number analyzed (Participants) | 0 | 29 | 25 | 14 | 18
  Week 4 |  | 17 | 10 | 9 | 5
  Week 8: number analyzed (Participants) | 0 | 28 | 22 | 13 | 17
  Week 8 |  | 17 | 10 | 9 | 4
  Week 12: number analyzed (Participants) | 0 | 27 | 21 | 13 | 15
  Week 12 |  | 20 | 10 | 9 | 5
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.2674, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.46 to 10.67] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.2850, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.78, 95% CI 2-sided [0.44 to 17.54] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.3086, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.63, 95% CI 2-sided [0.42 to 16.52] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 4: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.1655, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 4.33, 95% CI 2-sided [0.46 to 40.83] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 5: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.7154, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.26 to 7.67] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 6: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.5371, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.27 to 14.64] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 7: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.2170, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 5.00, 95% CI 2-sided [0.43 to 57.83] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 8: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.3408, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.41 to 18.22] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 9: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.3270, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.41 to 14.20] — Stratified by pooled site group and baseline IGA grade
Statistical Analysis 10: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.0719, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade
Statistical Analysis 11: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID; Week 12; Test type: Superiority; p = 0.8527, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.07 to 8.43]
Statistical Analysis 12: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.3545, Cochran-Mantel-Haenszel; Stratified by pooled site group and baseline IGA grade; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.37 to 13.11]

16. Secondary Outcome: Cohort 2: Change From Baseline in Overall Quality of Life in Hand Eczema Questionnaire (QOLHEQ) Score at Each Visit
Description: The QOLHEQ is an instrument to assess disease specific Health Related Quality of Life (HRQOL) in patients suffering from hand eczema. The QOLHEQ is a disease specific instrument, thereby only assessing impairments caused by hand eczema. It consists of 30 items which can be summarized according to four domains of HRQOL: Impairments because of (1) symptoms, (2) emotions, (3) limitations in functioning or (4) because of treatment and prevention. The scoring ranges from 0 ('no eczema') to 117 ('most severe eczema').
Time Frame: Weeks 2, 4, 8, 12, 13
Population: All participants in Cohort 2 with data available are included.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 62 | 59 | 30 | 63
score on a scale
  Week 2 |  | -13.7 (1.89) | -15.1 (1.92) | -11.0 (2.64) | -9.3 (1.86)
  Week 4: number analyzed (Participants) | 0 | 61 | 56 | 29 | 55
  Week 4 |  | -17.4 (2.44) | -18.5 (2.49) | -15.3 (3.45) | -13.4 (2.56)
  Week 8: number analyzed (Participants) | 0 | 56 | 54 | 27 | 51
  Week 8 |  | -16.6 (2.59) | -19.6 (2.61) | -20.8 (3.65) | -12.0 (2.67)
  Week 12: number analyzed (Participants) | 0 | 59 | 50 | 28 | 46
  Week 12 |  | -19.2 (2.77) | -24.9 (2.95) | -22.3 (3.89) | -15.3 (3.04)
  Week 13: number analyzed (Participants) | 0 | 59 | 49 | 27 | 46
  Week 13 |  | -20.9 (2.76) | -22.9 (2.89) | -18.9 (3.81) | -15.6 (3.04)
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.0725, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-9.2 to 0.4] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.0183, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-10.7 to -1.0] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.5701, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-7.7 to 4.3]
Statistical Analysis 4: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.2116, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-10.4 to 2.3] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 5: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.1235, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-11.5 to 1.4] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 6: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.6334, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-9.7 to 5.9] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 7: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.1788, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-11.4 to 2.1] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 8: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.0292, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -7.6, 95% CI 2-sided [-14.4 to -0.8] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 9: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.0371, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-17.1 to -0.5] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 10: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.2971, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-11.3 to 3.5] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 11: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.0150, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -9.5, 95% CI 2-sided [-17.2 to -1.9] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 12: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.1245, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-15.8 to 1.9] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 13: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 13; Test type: Superiority; p = 0.1591, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-12.7 to 2.1] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 14: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 13; Test type: Superiority; p = 0.0600, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-14.8 to 0.3] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 15: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 13; Test type: Superiority; p = 0.4640, ANCOVA; Treatment group, pooled site group, and baseline IGA were independent variables; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-12.0 to 5.5] — Treatment group, pooled site group, and baseline IGA were independent variables

17. Secondary Outcome: Cohort 2: Change From Baseline in Total Body Surface Area (BSA) Affected by Disease
Description: The percentage of total body surface area (BSA) affected by chronic hand eczema (CHE) is a measure of the area of the subject's hands that is affected by CHE lesions, expressed as a percentage of total BSA. Based on the subject's hand method, the BSA of 1 side of 1 hand is assumed to be 1% of total BSA. The surface area of lesions on both sides of both hands are added to calculate the total BSA affected by CHE. The total BSA affected by CHE ranges from 0% (no CHE lesions) to 4% (the entire front and back sides of both hands are affected by CHE lesions).
Time Frame: Weeks 2, 4, 8, 12
Population: All participants in Cohort 2 with data available are included.
Measure: Mean (Standard Error); unit: Percentage of Total BSA
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream Pooled
Number analyzed (Participants) | 0 | 61 | 52 | 31 | 63
Percentage of Total BSA
  Week 2 |  | -0.185 (0.0517) | -0.132 (0.0559) | -0.028 (0.0697) | -0.119 (0.0509)
  Week 4: number analyzed (Participants) | 0 | 60 | 50 | 29 | 54
  Week 4 |  | -0.310 (0.0583) | -0.319 (0.0634) | -0.151 (0.0818) | -0.139 (0.0616)
  Week 8: number analyzed (Participants) | 0 | 55 | 48 | 27 | 50
  Week 8 |  | -0.319 (0.0746) | -0.273 (0.0808) | -0.241 (0.1039) | -0.223 (0.0744)
  Week 12: number analyzed (Participants) | 0 | 58 | 46 | 28 | 45
  Week 12 |  | -0.429 (0.0681) | -0.409 (0.0759) | -0.296 (0.0948) | -0.307 (0.0751)
Statistical Analysis 1: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.3184, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.066, 95% CI 2-sided [-0.196 to 0.064] — Treatment group, pooled site group, and baseline IGA were independent variables
Statistical Analysis 2: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.8514, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.013, 95% CI 2-sided [-0.149 to 0.123] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 3: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 2; Test type: Superiority; p = 0.2603, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [-0.068 to 0.249] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 4: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.0273, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.171, 95% CI 2-sided [-0.323 to -0.019] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 5: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.0266, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.180, 95% CI 2-sided [-0.339 to -0.021] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 6: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 4; Test type: Superiority; p = 0.9023, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.196 to 0.173] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 7: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.3298, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.096, 95% CI 2-sided [-0.291 to 0.098] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 8: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.6205, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.050, 95% CI 2-sided [-0.251 to 0.150] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 9: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 8; Test type: Superiority; p = 0.8817, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.253 to 0.217] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 10: Comparison: Cohort 2: ARQ-252 Cream 0.3% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.1837, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.122, 95% CI 2-sided [-0.302 to 0.058] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 11: Comparison: Cohort 2: ARQ-252 Cream 0.3% BID vs Cohort 2: Vehicle Cream Pooled; Test type: Superiority; p = 0.2896, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = -0.102, 95% CI 2-sided [-0.293 to 0.088] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables
Statistical Analysis 12: Comparison: Cohort 2: ARQ-252 Cream 0.1% QD vs Cohort 2: Vehicle Cream Pooled; Week 12; Test type: Superiority; p = 0.9190, ANCOVA; Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.205 to 0.227] — Treatment group, pooled site group, baseline IGA grade, and baseline % BSA were independent variables

ADVERSE EVENTS:
Time Frame: Up to ~14 weeks
Description: All treated participants are included.
Arm/Group | Cohort 1: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% QD | Cohort 2: ARQ-252 Cream 0.3% BID | Cohort 2: ARQ-252 Cream 0.1% QD | Cohort 2: Vehicle Cream QD | Cohort 2: Vehicle Cream BID
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/65 | 0/61 | 0/32 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/65 | 0/61 | 0/32 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/7 | 2/65 | 2/61 | 3/32 | 2/33 | 1/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ARQ-252 Cream 0.3% QD (N=7) | Cohort 2: ARQ-252 Cream 0.3% QD (N=65) | Cohort 2: ARQ-252 Cream 0.3% BID (N=61) | Cohort 2: ARQ-252 Cream 0.1% QD (N=32) | Cohort 2: Vehicle Cream QD (N=33) | Cohort 2: Vehicle Cream BID (N=32)
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT04378569/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT04378569/SAP_001.pdf